CLINICAL TRIAL: NCT02491411
Title: A Pilot Study of Dexamethasone Therapy Prior to Rechallenge With Enzalutamide in Men With Metastatic Castration-Resistant Prostate Cancer Dex EXTends Enza Response (The DEXTER Trial)
Brief Title: Dexamethasone Prior to Re-treatment With Enzalutamide in Treating Patients With Metastatic Hormone-Resistant Prostate Cancer Previously Treated With Enzalutamide and Docetaxel
Acronym: DEXTER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study is terminated due to lower enrollment
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1548; NCI-2015-00918 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB00064598; J1548 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); P30CA006973 (NIH)
Record Dates: First submitted 2015-06-18; First posted 2015-07-08 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Hormone-Resistant Prostate Cancer; Metastatic Prostate Carcinoma; Prostate Adenocarcinoma; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (dexamethasone and enzalutamide) (Experimental): Patients receive dexamethasone PO once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity until there is evidence of PSA progression, clinical disease progression, or radiographic disease progression. At time of progression, dexamethasone will be stopped via a rapid taper over one week if patients were treated for over 30 days. Patients then receive enzalutamide PO once daily on days 1-28. Treatment repeats every 28 days for up to 3 courses in the absence of clinical disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Drug: Enzalutamide; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Enzalutamide — Given PO
  Other Names: MDV3100; Xtandi
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This pilot trial studies how well dexamethasone and re-treatment with enzalutamide work in treating patients with prostate cancer that has spread to other places in the body (metastatic), does not respond to hormone therapy (hormone-resistant), and was previously treated with enzalutamide and docetaxel. Dexamethasone treatment may be able to reverse one resistance mechanism to enzalutamide therapy (overabundance of receptors for dexamethasone and other glucocorticoids inside cancer cells) and allow for renewed therapeutic sensitivity to enzalutamide. Androgens (a type of male hormone) can bind to androgen receptors found inside prostate cancer cells, which may cause the cancer cells to grow. Enzalutamide may stop the growth of prostate cancer cells by blocking the activity of the cancer cell androgen receptors. Giving dexamethasone prior to re-treatment with enzalutamide may be a treatment for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the prostate-specific antigen (PSA) response rate to enzalutamide (Enza) after treatment with dexamethasone (Dex) therapy.

SECONDARY OBJECTIVES:

I. Objective response rate to Enza in patients with measurable disease on computed tomography (CT) scan using Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

II. Time to PSA progression (based upon Prostate Cancer Working Group 2 [PCWG2] criteria) for treatment with Dex.

III. Effect of each treatment on quality of life as assessed by patient completion of validated instruments (Functional Assessment of Chronic Illness Therapy [FACIT]-Fatigue Scale, RAND Short Form-36 [RANDSF-36]).

IV. PSA response rates to Dex for patients who are androgen receptor splice variant 7 (AR-V7) positive and AR-V7 negative, respectively, at study entry.

V. Response rates to Enza for patients who are AR-V7 positive and AR-V7 negative, respectively, at study entry.

VI. Percentage of patients who are AR-V7 positive at study entry who are AR-V7 negative at time of initiation of Enza, or vice-versa.

OUTLINE:

Patients receive dexamethasone orally (PO) once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity until there is evidence of PSA progression, clinical disease progression, or radiographic disease progression. At time of progression, dexamethasone will be stopped via a rapid taper over one week if patients were treated for over 30 days. Patients then receive enzalutamide PO once daily on days 1-28. Treatment repeats every 28 days for up to 3 courses in the absence of clinical disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma of the prostate
* Patients must have metastatic disease radiographically documented by CT/magnetic resonance imaging (MRI) or bone scan; measurable disease is not necessary for inclusion
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months in the opinion of the investigator
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 8; transfusion is allowed
* Total bilirubin =< 1.5 x institutional upper limit of normal
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine clearance >= 30 by Cockcroft-Gault formula
* Patients must have progression after prior treatment with Enza at any point in the disease course (pre- or post-chemotherapy)
* Patients must have progressed after prior treatment with docetaxel; docetaxel must have specifically been given for castration-resistant metastatic disease
* Prior treatment with other second line hormone therapy is allowed (e.g. flutamide, bicalutamide, nilutamide, ketoconazole, abiraterone, ARN-509); patients must be off these therapies for at least 4 weeks prior to starting treatment
* Prior treatment with Xofigo (223Radium), Provenge, mitoxantrone and cabazitaxel is allowed
* Patients must have rising PSA on two successive measurements, at least 2 weeks apart
* Patient must be treated with continuous androgen ablative therapy (e.g. goserelin, leuprolide, triptorelin, or degarelix, if he has not had prior surgical castration) and have castrate levels of testosterone (< 50 ng/dL or 1.7 nmol/L)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier (persistent toxicity >= grade 1)
* Patients who have received any other investigational agents within the last 4 weeks
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Dex or Enza
* Any use of systemic corticosteroids in the prior 4 weeks
* Uncontrolled diabetes mellitus
* History of seizure, underlying brain injury with loss of consciousness, transient ischemic attack within the past 12 months, cerebral vascular accident, brain metastases, and brain arteriovenous malformations
* Patients receiving any medications or substances that are inhibitors or inducers of cytochrome P450 family 2, subfamily C, polypeptide 8 (CYP2C8) are ineligible (e.g. gemfibrozil, rifampin, trimethoprim, pioglitazone)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations or geographical condition that would limit compliance with study requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Denmeade, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (1):
- Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One of the five patients enrolled, failed screen due to declining Eastern Cooperative Oncology Group (ECOG) Score of 3, and therefore could not start study.
Groups:
- Treatment (Dexamethasone and Enzalutamide): Patients receive dexamethasone PO once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity until there is evidence of prostate specific antigen (PSA) progression, clinical disease progression, or radiographic disease progression. At time of progression, dexamethasone will be stopped via a rapid taper over one week if patients were treated for over 30 days. Patients then receive enzalutamide PO once daily on days 1-28. Treatment repeats every 28 days for up to 3 courses in the absence of clinical disease progression or unacceptable toxicity.
  Dexamethasone: Given PO
  Enzalutamide: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Quality-of-Life Assessment: Ancillary studies
Period: Overall Study
Arm/Group | Treatment (Dexamethasone and Enzalutamide)
Started | 4
Completed | 0
Not Completed | 4
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Dexamethasone and Enzalutamide)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: PSA Response Rate
Description: PSA response rate is defined as the proportion of subjects with a >= 50% PSA decline from baseline level when starting enzalutamide and maintained for >= 4 weeks at any time-point after receiving enzalutamide. Will determine its corresponding 95% confidence interval.
Time Frame: Up to 4 weeks post-treatment
Population: Data was not collected, the study was terminated early due to lower enrollment.
Arm/Group | Treatment (Dexamethasone and Enzalutamide)
Number analyzed (Participants) | 0

2. Secondary Outcome: Changes in Quality of Life Assessment Scores, Assessed Using FACIT-Fatigue Scale and RANDSF-36 Surveys
Description: Summary statistics of the scores will be reported at baseline before starting dexamethasone and each follow-up time during the treatment of dexamethasone and enzalutamide. Changes in quality of life scores over the course of the study will be computed and their significance will be evaluated by paired-sample t-tests.
Time Frame: Baseline to up to 4 weeks post-treatment
Population: Data was not collected, the study was terminated early due to lower enrollment.
Arm/Group | Treatment (Dexamethasone and Enzalutamide)
Number analyzed (Participants) | 0

3. Secondary Outcome: Objective Response Rate to Enzalutamide in Patients With Measurable Disease on CT Scan
Description: Will estimate 95% confidence interval.
Time Frame: Up to 4 weeks post-treatment
Population: Data was not collected, the study was terminated early due to lower enrollment.
Arm/Group | Treatment (Dexamethasone and Enzalutamide)
Number analyzed (Participants) | 0

4. Secondary Outcome: Response Rate With Dexamethasone by AR-V7 Status at Study Entry
Time Frame: Baseline
Population: Data was not collected, the study was terminated early due to lower enrollment.
Arm/Group | Treatment (Dexamethasone and Enzalutamide)
Number analyzed (Participants) | 0

5. Secondary Outcome: Response Rate With Enzalutamide by AR-V7 Status at Study Entry
Time Frame: Baseline
Population: Data was not collected, the study was terminated early due to lower enrollment.
Arm/Group | Treatment (Dexamethasone and Enzalutamide)
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to PSA Progression, Based Upon PCWG2 Criteria, for Treatment With Dexamethasone
Description: Will be summarized using Kaplan-Meier approach.
Time Frame: Up to 4 weeks post-treatment
Population: Data was not collected, the study was terminated early due to lower enrollment.
Arm/Group | Treatment (Dexamethasone and Enzalutamide)
Number analyzed (Participants) | 0

7. Secondary Outcome: Time to Radiographic Progression for Treatment With Dexamethasone
Description: Will be summarized using Kaplan-Meier approach.
Time Frame: Up to 4 weeks post-treatment
Population: Data was not collected, the study was terminated early due to lower enrollment.
Arm/Group | Treatment (Dexamethasone and Enzalutamide)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 weeks post treatment for each treatment cycle, up to 1 year
Description: Every visit
Arm/Group | Treatment (Dexamethasone and Enzalutamide)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Dexamethasone and Enzalutamide) (N=4)
cushingoid (increased appetite and weight ) (Endocrine disorders) | 2 (2)
insomnia (Nervous system disorders) | 2 (2)
left hand cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
irritability (Nervous system disorders) | 1 (1)
fatigue (General disorders) | 2 (2)
abdominal pain (General disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
BILATERAL LOWER EXTREMITIES EDEMA (Skin and subcutaneous tissue disorders) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Paresthesia (Investigations) | 1 (1)
Right rib pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Eye disorders (reddened eyes) (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-08-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT02491411/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT02491411/SAP_001.pdf